CLINICAL TRIAL: NCT05029154
Title: Effect of Exercise Preconditioning in Ovarian Cancer on Treatment-Related Cardiotoxicity
Brief Title: Exercise Preconditioning in Ovarian Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual not meeting pre-specified numbers.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Siddartha Angadi, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSR210169
Record Dates: First submitted 2021-08-17; First posted 2021-08-31 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer
Keywords: Cardiotoxicity; Ovarian Cancer; Exercise Training; Chemotherapy; Cardiovascular toxicity ovarian cancer chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Cardiotoxicity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Two-arm randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention (i.e. exercise training), participants and study team members cannot be blinded. However, outcomes assessment will be carried out in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients in the exercise group will perform interval training 3 days per week.
  Interventions: Behavioral: High intensity interval exercise
- Attention Control (Placebo Comparator): Physical activity education and physical activity monitoring.
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: High intensity interval exercise — Patients in the exercise group will perform interval training (HIIT) 3 days per week, with each session consisting of four, 4-min intervals at 85-90% peak heart rate (PHR), separated by 3 min at 50% PHR. Each training session will begin with a 10-minute warm-up at 50% of PHR and end with a 5-min cool down at 50% PHR. Patients will undergo 2 initial training sessions at the exercise physiology core lab. All exercise will consist of stationary cycling to avoid discomfort associated with abdominal surgery as well as stress to the incision and help reduce fall risk. Study investigators will check in weekly with participants and remotely track exercise data and compliance via the Fitbit app.
  Arms: Exercise
Behavioral: Attention control — Patients in the control group (physical activity education and physical activity monitoring) will receive counseling regarding the benefits of physical activity during chemotherapy treatment. During the intervention, participants will receive a weekly phone call to discuss their physical activity and remind them to engage in physical activity. Patients will be given a goal of working up to 30 minutes of exercise daily. Subjects will be urged to increase daily step counts by 250-500 steps/day. Physical activity will be objectively assessed and made available to the participant using a Fitbit.
  Arms: Attention Control

SUMMARY:
The purpose of this study is to determine if exercise preconditioning can mitigate the off target effects of chemotherapy treatment on measures of cardiovascular function, peripheral neuropathy, and quality of life.

DETAILED DESCRIPTION:
While survivorship for those diagnosed with epithelial ovarian cancer has continued to improve, the significant off target effects of adjuvant and neoadjuvant chemotherapy have become more prominent. These off-target effects include increased risk of cardiovascular disease, neuropathy, and decreased quality of life. Exercise initiated prior to chemotherapy induction and continued through treatment has promise in terms of preserving VO2peak and potentially mitigating the negative cardiovascular and neuropathic effects of chemotherapy. The goal of this study is to examine the effects of initiating exercise prior to any oncologic therapy and sustaining this exercise paradigm in newly diagnosed women with ovarian cancer who are undergoing initial surgery and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Presumed diagnosis of ovarian cancer and a planned chemotherapy regimen of a taxane and carboplatin with or without VEGF inhibition
* Physician clearance for exercise training

Exclusion Criteria:

* Any patient unable/unwilling to cooperate with all study protocols
* Cancer recurrence
* Previous treatment with chemotherapy in the last 5-years
* Medical/orthopedic co-morbidities that preclude exercise training
* Significant heart, liver, kidney, blood, or respiratory disease precluding exercise participation
* Peripheral vascular disease
* Acute infectious disease or history of chronic infections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
VO2 Peak | 22 weeks
  Change in VO2peak (L/min) measured at pre-surgery, pre-chemotherapy, and post chemotherapy

SECONDARY OUTCOMES:
Global Longitudinal Strain | 22 weeks
  Global longitudinal strain (%) will be used to assess changes in cardiac contractile function and be measured by echocardiogram at pre-surgery, pre-chemotherapy, and post-chemotherapy
Ejection Fraction | 22 weeks
  Ejection fraction (%) will be used to assess changes in cardiac contractile function and be measured by echocardiogram at pre-surgery, pre-chemotherapy, and post-chemotherapy
Diastolic Function | 22 weeks
  E' and A' (cm/s) will be used to calculate the E'/A' ratio to assess for diastolic dysfunction and be measured by echocardiogram at pre-surgery, pre-chemotherapy, and post-chemotherapy
Brachial Artery Endothelium-Dependent Flow-Mediated Dilation | 22 weeks
  Changes in endothelial function as measured by brachial artery endothelium-dependent flow-mediated dilation (%) at pre-surgery, pre-chemotherapy, and post-chemotherapy
Carotid-Femoral Pulse Wave Velocity | 22 weeks
  Changes in arterial stiffness as measured by carotid-femoral pulse wave velocity (m/s) at pre-surgery, pre-chemotherapy, and post-chemotherapy
Blood pressure | 22 weeks
  Changes in measures of central and brachial blood pressure (mmHg) at pre-surgery, pre-chemotherapy, and post-chemotherapy
Peripheral Neuropathy | 22 weeks
  A Neuropen will be used to assess for peripheral neuropathy via changes in perception to pressure prior to chemotherapy, at cycle 4, and after cycle 6.
Peripheral Neuropathy as assessed by the FACT-GOG-NTX Questionnaire | 22 weeks
  The functional assessment of cancer therapy/gynecologic oncology group- neurotoxicity (FACT-GOG-NTX) questionnaire is used to assess symptoms of peripheral neuropathy. This 38 item questionnaire utilizes the same questions as the FACT questionnaire with 11 questions specific to peripheral neuropathy. A 5 point Likert scale is used for each question and subscores are added together with high scores indicating better quality of life
Health Related Quality of Life as Measured by the FACT-O Questionnaire | 22 weeks
  The functional assessment of cancer therapy- ovarian cancer(FACT-O) questionnaire is used to assess health-related quality of life specific to cancer and includes a subscale for ovarian cancer. This 38 item questionnaire utilizes the same questions as the FACT questionnaire with 12 questions specific to ovarian cancer. A 5 point Likert scale is used for each question and subscores are added together with high scores indicating better quality of life
Quality of Life as Assessed by the Short Form Health Survey (SF-36) | 22 weeks
  The Short Form Health survey is a 36 item questionnaire that is used to measure general health and quality of life. Responses in each section are scored on a scale of 0-100 (with 100 indicating good health) and averaged together for each subscale score.

OTHER OUTCOMES:
NTproBNP | 22 weeks
  Assess changes in NTproBNP (pg/ml) as a biomarker of myocardial strain at pre-surgery, pre-chemotherapy, and post-chemotherapy
Inflammation | 22 weeks
  C-reactive protein (mg/dl) will be used as a biomarker for inflammation to be measured at pre-surgery, pre-chemotherapy, and post-chemotherapy
Lipids | 22 weeks
  A lipid panel will be performed to measure total cholesterol, triglycerides, high-density lipoproteins, and low-density lipoprotein (mg/dl) to assess changes in cardiometabolic health at pre-surgery, pre-chemotherapy, and post-chemotherapy
Insulin | 22 weeks
  Fasting insulin levels (U/ml) will be tested to assess changes in cardiometabolic health at all 3 time points
Fasting Blood Glucose | 22 weeks
  Fasting blood glucose levels (mg/dl) will be tested to assess changes in cardiometabolic health at pre-surgery, pre-chemotherapy, and post-chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha S Angadi, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia University Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No